CLINICAL TRIAL: NCT00327080
Title: Evaluation of Endothelial and Hemodynamic Function in HIV Associated Pulmonary Hypertension and a Phase I/II Safety and Efficacy Trial of Sildenafil in HIV Associated Pulmonary Hypertension
Brief Title: Sildenafil to Treat HIV-Associated Pulmonary Hypertension
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060165; 06-H-0165
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2012-11-13

CONDITIONS: HIV
Keywords: HIV; AIDS; Pulmonary Hypertension; Blood Flow Studies; Right Heart Catheterization; HIV Infection; HIV Associated Pulmonary Hypertension; Healthy Volunteer; HV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hypertension, Pulmonary; HIV Infections | interventions — omega-N-Methylarginine; Acetylcholine

INTERVENTIONS:
Procedure: MRI
Drug: L-NMMA
Drug: Acetylcholine

SUMMARY:
This study will examine how blood pressure in the lungs is controlled in healthy people, people with HIV and people with HIV and pulmonary artery hypertension (high blood pressure in the lungs, also called PAH). PAH sometimes develops in people with HIV, but it is not known why this occurs or how best to treat it.

Healthy volunteers and patients with HIV infection who are 18 years of age or older may be eligible for this study. All candidates are screened with a medical history, physical examination, electrocardiogram (EKG), chest x-ray, echocardiogram and blood tests. Participants undergo the following procedures:

All participants have a right heart catheterization and forearm blood flow study.

* Catheterization study. A catheter (plastic tube) is placed in an arm vein and possibly in an artery in the arm. Then a large catheter is passed through a vein in the groin, neck or chest. Through this "introducer" catheter, another catheter is advanced into the right side of the heart and to the pulmonary artery. A facemask is put in place to measure the amount of nitric oxide produced by the lungs. Acetylcholine is infused through the catheter and its effects on blood pressure in the lungs and on the amount of nitric oxide exhaled is measured. After about 1 hour, the catheter and facemask are removed and a new catheter is inserted through the introducer catheter into the pulmonary artery. The subject is moved into an MRI scanner where blood flow is measured after infusion of three different medications: acetylcholine (causes blood vessels to expand and slows heart rate); sodium nitroprusside (causes blood vessels to expand and increases blood flow to the heart); and L-NMMA (decreases blood flow by blocking production of nitric oxide in cells lining the blood vessels).
* Blood flow study. Small tubes are inserted into the artery of the patient's forearm. These are used to infuse medicines and draw blood samples. Forearm blood flow is measured using pressure cuffs placed on the wrist and upper arm, and a strain gauge (a rubber band device) placed around the forearm. When the cuffs are inflated, blood flows into the arm, stretching the strain gauge, and the flow measurement is recorded. A small lamp is positioned over the hand to measure the light reflected from the hand and blood flow in the forearm. Blood samples are then drawn to measure blood counts and proteins and other natural body chemicals. Then, forearm blood flow is measured after administration of small doses of sodium nitroprusside, acetylcholine and L-NMMA. There is a 20- to 30-minute rest period between injections of the different drugs.

In addition, HIV-infected patients with PAH undergo the following tests to determine the cause of their PAH: CT scan of the lungs, pulmonary function tests, 6-minute walk test, quality-of-life assessment, assessment of difficulty in breathing, exercise testing while measuring oxygen breathed in and carbon dioxide breathed out, blood tests, monitoring of oxygen saturation during sleep for 1 night and ventilation/perfusion scan. For the ventilation/perfusion scan, the subject breathes in a small amount of radioactive aerosol while images are obtained of the radioactivity as it enters the lungs, and then pictures of the lungs are taken from multiple angles. Next, the patient receives an injection of tiny particles of albumin (a protein) containing a small amount of radioactivity and pictures of the lungs are taken that show the pattern of blood flow to the lungs.

Patients with HIV and PAH who may benefit from the investigational drug, sildenafil (commonly known as Viagra), may continue to participate in the next stage of the study. They receive the first dose of sildenafil after completing the forearm blood flow study. They continue the drug for 16 weeks, returning to the clinic 1 week after the first dose and then every other week to monitor the response to treatment and drug side effects. At the end of 16 weeks, patients return to the clinic for a repeat evaluation, including blood tests, 6-minute walk test, echocardiogram, right heart catheterization and forearm blood flow study.

...

DETAILED DESCRIPTION:
HIV infection has been associated with an increased prevalence of pulmonary hypertension. In addition, recent data suggests that a state of endothelial dysfunction develops in HIV disease secondary to anti-retroviral therapy and associated dyslipidemia or secondary to direct viral infection of the endothelium. This leads to premature atherosclerosis and possibly contributes to avascular necrosis of the hip. Similar effects on the pulmonary vasculature may be involved in the development of pulmonary vasculopathy.

In this study we plan to invasively characterize the status of pulmonary and systemic endothelial function and determine the mechanisms of pulmonary vascular endothelial dysfunction in HIV disease. To this end we will catheterize healthy volunteers and volunteers with HIV infection with and without pulmonary hypertension and directly measure acetylcholine-dependent blood flow in the pulmonary and brachial artery to assess pulmonary and systemic endothelium-dependent blood flow. Simultaneous measurement of exhaled NO and pulmonary capillary artery NO2 - will allow for complete characterization of the contribution of NO production to endothelium-dependent vasomotor control. We will also use recently developed MRI techniques to measure pulmonary artery blood flow during infusion of acetylcholine (ACH), sodium nitroprusside (SNP) and NG monomethyl-L-arginine (LNMMA) to establish responsiveness to an endothelium dependent vasodilator, endothelium-independent vasodilator and an NO inhibitor, respectively. Volunteers with pulmonary hypertension will have the option to undergo open label phase I/II treatment with sildenafil for 16 weeks and return for a repeat assessment of pulmonary hemodynamics as well as pulmonary and systemic endothelial function.

Endothelial cells will be isolated using novel flow-cytometry methodologies developed over the last two years at the NIH intramural division utilizing combinations of positive and negative selection based on specific surface markers for activated T cells and endothelial cells and markers of cell viability. Endothelial cells will subsequently be interrogated using amplified real time PCR methodologies and affymetrix based gene expression profiling developed in our laboratories. The levels of expression in endothelial cells of HIV virus, HHV8, eNOS, caveolin, HO-1, endothelin receptors A and B, and endothelin 1, in addition to other proteins regulating vascular homeostasis and cellular host defense (i.e. epidermal growth factor, transforming growth factor beta, platelet derived growth factor and interleukin-6), will be assessed.

These studies will provide insights into the mechanisms of pulmonary artery endothelial dysfunction and suggest rationally designed therapies targeting viral load, HHV8, and/or the NO/endothelin pathways. These studies have the promise of opening the door to the study of pulmonary artery endothelial dysfunction at the physiological, cellular and molecular level.

ELIGIBILITY:
* INCLUSION CRITERIA:

All volunteer subjects must be at least 18 years of age and must be able to provide informed, written consent for participation in this study. Eligibility in the study is determined prior to enrollment on the basis of the following inclusion and exclusion criteria.

For Healthy Volunteers:

1. Males or females, 18 years of age or older.
2. No history of HIV infection.
3. EKG and echocardiogram with no evidence of clinical relevant heart disease (including TRV less than 2.5 m/s)
4. No history of causes of pulmonary hypertension such as collagen vascular disease, chronic liver disease with ALT or AST greater than 2 times the upper limit of normal or cirrhosis of the liver, chronic thromboembolic disease, congenital heart defects, or pulmonary parenchymal disease with hypoxemia.
5. No history of diseases thought to be related to development of endothelial dysfunction including systemic hypertension or diabetes requiring drug therapy, hypercholesterolemia and obesity.
6. No history of anemia, thrombocytopenia or coagulopathy.
7. No history of renal insufficiency.
8. No medical conditions requiring chronic medication use with the exception of:

   1. Heartburn, GERD
   2. Environmental allegeries, post nasal drip or non-allergic rhinitis
   3. Asthma with no history of oral steroid use, weekly inhaled steroids, or hospitalization for asthma exacerbation.
   4. Dermatologic conditions that do not require the use of oral steroids or other immunosuppressants.
9. No more than 20 cigarettes per year for the previous 2 years and no cigarette use for 30 days prior to the screening evaluation until completion of the study.

For HIV Positive Volunteers:

1. Males or females, 18 years of age or older.
2. Diagnosis of HIV infection.
3. Under the care of a primary care physician.
4. No history of other potential causes of pulmonary hypertension such as collagen vascular disease, chronic liver disease with ALT or AST greater than 2 times the upper limit of normal or cirrhosis of the liver, chronic thromboembolic disease, congenital heart defects, or pulmonary parenchymal disease with hypoxemia.
5. For stage 3 enrollment: symptomatic pulmonary hypertension with MPAP greater than or equal to 25 mmHg and six-minute walk distance between 150-450 m.

EXCLUSION CRITERIA:

For Healthy volunteers:

1. Current pregnancy, lactation or women not currently using medically acceptable birth control. (All women of childbearing age will be required to have a screening urine or blood pregnancy test)
2. Contraindication to MRI scanning including individuals with the following devices:

   A) Central nervous system aneurysm clips

   B) Implanted neural stimulator

   C) Implanted cardiac pacemaker or defibrillator prior to enrollment

   D) Cochlear implant

   E) Ocular foreign body (e.g. metal shavings)

   F) Insulin pump

   G) Metal shrapnel or bullet
3. Contraindications to MRI contrast agent administration:
4. Inability to provide informed written consent for participation in the study.
5. Chronic, medically refractory atrial tachyarrhythmias
6. Symptoms of heart failure
7. Mean PA greater than 25 mmHg or PVR greater than 1.5 wood units, or PCWP greater than 15 mmHg
8. History of recreational drug use with the exception of marijuana. No Marijuana use within 3 months of protocol screening through completion of the study.

Volunteers may be excluded if in the opinion of the study investigators they have a condition that may adversely affect the outcome of the study or the safety of the volunteer.

For HIV Positive Volunteers:

1. Current pregnancy, lactation or women not currently using medically acceptable birth control.
2. Active, untreated opportunistic infection with the exception of oral thrush or neoplasm with the exception of Kaposi's Sarcoma.
3. Any of the following medical conditions:

   A) Severe renal insufficiency (on hemodialysis or serum creatinine greater than 2.5 mg/dl) or (CrCl less than 20 ml/min).

   B) Severe coagulopathy (platelets less than 100,000, PT INR greater than 1.5, PTT greater than 40 s)
4. Chronic, medically refractory atrial tachyarrhythmias
5. Current recreational drug use or use within 4 weeks of protocol screening with the exception of marijuana
6. Contraindication to MRI scanning including individuals with the following devices:

   A) Central nervous system aneurysm clips

   B) Implanted neural stimulator

   C) Implanted cardiac pacemaker or defibrillator prior to enrollment

   D) Cochlear implant

   E) Ocular foreign body (e.g. metal shavings)

   F) Insulin pump

   G) Metal shrapnel or bullet
7. Contraindications to MRI contrast agent administration:

A) Individuals with hemoglobinopathies

Volunteers may be excluded if in the opinion of the study investigators they have a condition that may adversely affect the outcome of the study or the safety of the volunteer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-05-12; Primary Completion 2009-03-18 (Actual); Study Completion 2009-03-18 (Actual)

PRIMARY OUTCOMES:
Evaluate pulmonary artery and systemic endothelial function in HIV infected volunteers with pulmonary hypertension in comparison to HIV infected volunteers without pulmonary hypertension.

SECONDARY OUTCOMES:
Evaluate the safety and efficacy of sildenafil in the treatment of hemodynamic and functional abnormalities in volunteers with HIV associated pulmonary hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Masur, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Opravil M, Pechere M, Speich R, Joller-Jemelka HI, Jenni R, Russi EW, Hirschel B, Luthy R. HIV-associated primary pulmonary hypertension. A case control study. Swiss HIV Cohort Study. Am J Respir Crit Care Med. 1997 Mar;155(3):990-5. doi: 10.1164/ajrccm.155.3.9117037.
- [Background] Zuber JP, Calmy A, Evison JM, Hasse B, Schiffer V, Wagels T, Nuesch R, Magenta L, Ledergerber B, Jenni R, Speich R, Opravil M; Swiss HIV Cohort Study Group. Pulmonary arterial hypertension related to HIV infection: improved hemodynamics and survival associated with antiretroviral therapy. Clin Infect Dis. 2004 Apr 15;38(8):1178-85. doi: 10.1086/383037. Epub 2004 Apr 1. PMID 15095226
- [Background] Nunes H, Humbert M, Sitbon O, Morse JH, Deng Z, Knowles JA, Le Gall C, Parent F, Garcia G, Herve P, Barst RJ, Simonneau G. Prognostic factors for survival in human immunodeficiency virus-associated pulmonary arterial hypertension. Am J Respir Crit Care Med. 2003 May 15;167(10):1433-9. doi: 10.1164/rccm.200204-330OC. Epub 2003 Feb 25. PMID 12615632